CLINICAL TRIAL: NCT01772329
Title: Preoperative Cognitive Therapy for Improving Health Outcomes After Total Knee Replacement in High-risk Catastrophizing Subjects
Brief Title: Preoperative Cognitive Therapy for Improving Health Outcomes After TKA in High-risk Catastrophizing Subjects
Acronym: CT_TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Profesor Anesthesiology, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12031901
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Catastrophization
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: n=80 Subjects for Aim 1 and another n=80 Subjects for Aim 2
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4 weekly CT sessions - in person (Experimental): 4 weekly CT sessions; all will be 1-hr individual cognitive therapy sessions with the psychology staff (under the supervision of John Burns, PhD).
  Interventions: Other: Cognitive Therapy
- 8 weekly CT sessions (Experimental): 8 weekly CT sessions; 1st and 8th will be 1-hr individual cognitive therapy session with the psychology staff (under the supervision of John Burns, PhD). The intermediate CT sessions will be by telephone call or video/"Skype". Our group will purchase and setup a web camera and headphone/microphone for the subjects in the CT groups that use "Skype". The 1-hr CT protocol was adapted from Dr. Beverly E. Thorn's CT manual (Cognitive Therapy for Chronic Pain: A Step-by-Step Guide; Thorn, 2004; with the Client and Therapy Workbooks.
  Interventions: Other: Cognitive Therapy
- 4 weekly CT sessions - Tele-video (Experimental): 4 weekly CT sessions; 1st and 4th will be 1-hr individual cognitive therapy session with the psychology staff. The intermediate CT sessions will be by telephone call or video/"Skype".
  Interventions: Other: Cognitive Therapy
- Routine care (Placebo Comparator): Routine care; no CT sessions
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Cognitive Therapy — CT will be used as a preemptive treatment in an effort to minimize the effects of catastrophic thinking.
  Arms: 4 weekly CT sessions - Tele-video; 4 weekly CT sessions - in person; 8 weekly CT sessions
Other: Routine Care — Routine Care. No Cognitive Therapy Intervention
  Arms: Routine care

SUMMARY:
The investigators propose a randomized controlled trial to evaluate the effects of treatment intended to reduce pain catastrophizing among patients reporting high pain catastrophizing prior to total knee replacement(TKR), total hip replacement(THR), or shoulder surgery in an effort to thereby reduce the incidence of persistent post-surgical pain (PPP) and enhance physical function at 3-months post-surgery. Preemptive treatment aimed at a known predictor of PPP following total knee replacement is highly innovative and have potentially high impact for public health. Cognitive therapy is a well-tolerated modality among chronic pain patients with few if any side effects. Cognitive therapy (CT) represents an inexpensive method that could greatly reduce suffering and costly post-surgical pain management for high risk TKR patients.

DETAILED DESCRIPTION:
Aim 1 is to determine which CT protocol is most effective in reducing Pain Catastrophizing Scale (PCS) and Coping Strategies Questionnaire Catastrophizing Subscale (CSQ-CAT) scores in high-risk TKR candidates. CT will consist of four-to-eight weekly 1-hr individual cognitive therapy sessions prior to surgery.

Aim 2 is to compare the most efficient treatment from Aim 1 with a control group to evaluate pain relief at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing standard primary TKR; THR or Shoulder Surgery
2. 18- 85 yrs of age;
3. Surgical joint is the primary source of patient's pain;
4. Patient agrees to preoperative visits and treatment, follow-up visits and treatment, and to comply with the assessment tests;
5. Patient consents to standard anesthetic and analgesic protocol, with medical care as deemed necessary by the anesthesiologist, and has no contraindications.
6. Patient has been diagnosed with osteoarthritis.

Exclusion Criteria:

1. Currently using antidepressant medication or undergoing cognitive therapy;
2. chronic opioid use ≥ 10 mg/day of morphine equivalents within one wk prior to the surgery, and duration of use > 4 wks;
3. history of opioid abuse;
4. inability to understand and communicate with the investigators to complete the study related questionnaires
5. patient is planning to undergo another elective joint procedure during the 6-mo period of participation;
6. any co-morbidity which results in severe systemic disease limiting function {as defined by the American Society of Anesthesiology (ASA) physical status classification > 3}.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
(Aim 1) Pain Catastrophizing Scale (PCS) | 4 or 8 weeks after start of treatment
  Pain Catastrophizing Scale - Min=0, Max=52, Higher score = more catastrophizing so lower scores are preferable.
(Aim 2) Proportion of patients with pain relief | 3 month
  Proportion of patients w a 3 month decrease in WOMAC pain subscale <= 4. (WOMAC Osteoarthritis Index)

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | 4 and 8 weeks after start of treatment
  Patient Health Questionnaire (PHQ-8): The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders
Generalized anxiety disorder (GAD-7) | 4 and 8 weeks after start of treatment
  Generalized anxiety disorder (GAD-7): The seven-item Generalized Anxiety Disorder Scale (GAD-7) is a practical self-report anxiety questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush UMC
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data as of yet but may be willing to.

REFERENCES:
- [Derived] Buvanendran A, Sremac AC, Merriman PA, Della Valle CJ, Burns JW, McCarthy RJ. Preoperative cognitive-behavioral therapy for reducing pain catastrophizing and improving pain outcomes after total knee replacement: a randomized clinical trial. Reg Anesth Pain Med. 2021 Apr;46(4):313-321. doi: 10.1136/rapm-2020-102258. Epub 2021 Jan 15. PMID 33452201